CLINICAL TRIAL: NCT00005676
Title: High Density Lipoprotein Subspecies and Coronary Disease
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bela Asztalos, Associate Professor, Tufts University
Other Study IDs: 909; R01HL064738 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Coronary Arteriosclerosis; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VA-HIT and FOS: VA-HIT cohort: men with established CHD and low HDL-C FOS cohort: men without CHD

SUMMARY:
To investigate the relative contributions of high density lipoprotein-C (HDL-C) subspecies to risk for coronary heart disease (CHD) in two distinct existing populations (samples from the VA-HIT study and the Framingham Offspring Study [FOS]) as well as the response of these subfractions to gemfibrozil treatment.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) continues to be a leading cause of death and disability in the United States. Information about the contribution of different subspecies of HDL-C to increased or decreased risk for premature CHD and the extent to which common lipoprotein lipase (LPL) mutations affect HDL-C composition and subspecies could contribute to an increased understanding of the role of HDL-C in determining CHD risk.

DESIGN NARRATIVE:

The following parameters will be measured in blood samples collected from the VA-HIT study and the Framingham Offspring Study: apo A-I-containing HDL subspecies (prebeta, alpha, and prealpha) in plasma using two-dimensional gel electrophoresis immunoblot and image analysis, LpA-I and LpA-I/A-II in plasma using differential electroimmunoassay, and apo C-III in HDL using immunoturbidometric assay. The study hypotheses are as follow. a) Subjects from the placebo arm of VA-HIT will have significantly lower alpha l HDL subspecies, LpA-I, and apo C-III in HDL, and higher HDL/alpha l and apo A-I/alpha l ratios than subjects free of coronary heart disease from the Framingham Offspring Study. b) These parameters will also predict prospectively risk of coronary heart disease in both groups. c) In the VA-HIT study, treatment with gemfibrozil, which has been shown to be associated with a 22 percent reduction in myocardial infarction and coronary heart disease death, will be associated with increases in alpha l HDL subspecies, LpA-I, and apo C-III in HDL, as well as decreases in HDL/alpha l and apo A-I/alpha l ratios, compared to placebo. d) The hypothesis that subjects with specific mutations in the lipoprotein lipase gene have less beneficial changes in HDL subspecies with gemfibrozil than subjects with no mutations will also be tested.

ELIGIBILITY:
VA-HIT: men, established CHD, HDL-C<40 mg/dl, LDL-C < 140 mg/dl, TG < 300 mg/dl FOS: men having no evidence of CHD

Ages: 41 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men with CHD and low HDL-C men without CHD
Sampling Method: Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2000-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
HDL subspecies | 1992-1998

CONTACTS AND LOCATIONS:
Overall Officials: Bela Asztalos, PhD, Principal Investigator — Tufts University

REFERENCES:
- [Background] Asztalos BF, Horvath KV, McNamara JR, Roheim PS, Rubinstein JJ, Schaefer EJ. Effects of atorvastatin on the HDL subpopulation profile of coronary heart disease patients. J Lipid Res. 2002 Oct;43(10):1701-7. doi: 10.1194/jlr.m200037-jlr200. PMID 12364554
- [Background] Asztalos BF, Brousseau ME, McNamara JR, Horvath KV, Roheim PS, Schaefer EJ. Subpopulations of high density lipoproteins in homozygous and heterozygous Tangier disease. Atherosclerosis. 2001 May;156(1):217-25. doi: 10.1016/s0021-9150(00)00643-2. PMID 11369017
- [Background] Lamon-Fava S, Posfai B, Asztalos BF, Horvath KV, Dallal GE, Schaefer EJ. Effects of estrogen and medroxyprogesterone acetate on subpopulations of triglyceride-rich lipoproteins and high-density lipoproteins. Metabolism. 2003 Oct;52(10):1330-6. doi: 10.1016/s0026-0495(03)00276-2. PMID 14564686
- [Background] Asztalos BF, Horvath KV, McNamara JR, Roheim PS, Rubinstein JJ, Schaefer EJ. Comparing the effects of five different statins on the HDL subpopulation profiles of coronary heart disease patients. Atherosclerosis. 2002 Oct;164(2):361-9. doi: 10.1016/s0021-9150(02)00149-1. PMID 12204809
- [Background] Asztalos BF, Batista M, Horvath KV, Cox CE, Dallal GE, Morse JS, Brown GB, Schaefer EJ. Change in alpha1 HDL concentration predicts progression in coronary artery stenosis. Arterioscler Thromb Vasc Biol. 2003 May 1;23(5):847-52. doi: 10.1161/01.ATV.0000066133.32063.BB. Epub 2003 Mar 13. PMID 12637338
- [Background] Asztalos BF, Cupples LA, Demissie S, Horvath KV, Cox CE, Batista MC, Schaefer EJ. High-density lipoprotein subpopulation profile and coronary heart disease prevalence in male participants of the Framingham Offspring Study. Arterioscler Thromb Vasc Biol. 2004 Nov;24(11):2181-7. doi: 10.1161/01.ATV.0000146325.93749.a8. Epub 2004 Sep 23. PMID 15388521
- [Background] Batista MC, Welty FK, Diffenderfer MR, Sarnak MJ, Schaefer EJ, Lamon-Fava S, Asztalos BF, Dolnikowski GG, Brousseau ME, Marsh JB. Apolipoprotein A-I, B-100, and B-48 metabolism in subjects with chronic kidney disease, obesity, and the metabolic syndrome. Metabolism. 2004 Oct;53(10):1255-61. doi: 10.1016/j.metabol.2004.05.001. PMID 15375779
- [Background] Asztalos BF; HDL Atherosclerosis Treatment Study. High-density lipoprotein metabolism and progression of atherosclerosis: new insights from the HDL Atherosclerosis Treatment Study. Curr Opin Cardiol. 2004 Jul;19(4):385-91. doi: 10.1097/01.hco.0000126979.41946.7e. PMID 15218401
- [Background] Yancey PG, Asztalos BF, Stettler N, Piccoli D, Williams DL, Connelly MA, Rothblat GH. SR-BI- and ABCA1-mediated cholesterol efflux to serum from patients with Alagille syndrome. J Lipid Res. 2004 Sep;45(9):1724-32. doi: 10.1194/jlr.M400133-JLR200. Epub 2004 Jun 21. PMID 15210845
- [Background] Webb NR, de Beer MC, Asztalos BF, Whitaker N, van der Westhuyzen DR, de Beer FC. Remodeling of HDL remnants generated by scavenger receptor class B type I. J Lipid Res. 2004 Sep;45(9):1666-73. doi: 10.1194/jlr.M400026-JLR200. Epub 2004 Jun 21. PMID 15210842
- [Background] Asztalos BF, Horvath KV, Kajinami K, Nartsupha C, Cox CE, Batista M, Schaefer EJ, Inazu A, Mabuchi H. Apolipoprotein composition of HDL in cholesteryl ester transfer protein deficiency. J Lipid Res. 2004 Mar;45(3):448-55. doi: 10.1194/jlr.M300198-JLR200. Epub 2003 Dec 1. PMID 14657195